CLINICAL TRIAL: NCT06227260
Title: Development and Evaluation of Body Massage Oil, Facial Mask, and Ready-to-drink Jelly From Snake Fruit (Salacca Edulis Reinw.)
Brief Title: Body Massage Oil, Facial Mask, and Ready-to-drink Jelly From Snake Fruit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burapha University (Other)
Responsible Party: Principal Investigator, Piyapong Prasertsri, Associate Professor Dr., Burapha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB1-028/2566
Record Dates: First submitted 2023-12-21; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Body Massage Oil From Snake Fruit; Facial Mask From Snake Fruit; Jelly From Snake Fruit
MeSH Terms: interventions — Medicine, Thai Traditional; Gels

STUDY DESIGN:
Intervention Model Description: Study 1 and 2 were parallel model, study 3 was crossover model.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Study 1: Thai massage (Active Comparator): Participants were randomized to receive an arm. In this arm, participants received Thai massage without any oil for 1 hour/day, 1 day/week for 12 weeks. Massage was performed at Burapha University by an expert.
  Interventions: Other: Thai massage, Thai massage with pure coconut oil, Thai massage with oil mixed with Snake fruit extract, Control, Facial mask with Snake fruit extract, Control jelly, Jelly with Snake fruit juice
- Study 1: Thai massage with pure coconut oil (Active Comparator): Participants were randomized to receive an arm. In this arm, participants received Thai massage with pure coconut oil which is a popular oil used in spa for 1 hour/day, 1 day/week for 12 weeks. Massage was performed at Burapha University by an expert.
  Interventions: Other: Thai massage, Thai massage with pure coconut oil, Thai massage with oil mixed with Snake fruit extract, Control, Facial mask with Snake fruit extract, Control jelly, Jelly with Snake fruit juice
- Study 1: Thai massage with oil mixed with Snake fruit extract (Experimental): Participants were randomized to receive an arm. In this arm, participants received Thai massage with oil mixed with Snake fruit extract for 1 hour/day, 1 day/week for 12 weeks. Massage was performed at Burapha University by an expert.
  Interventions: Other: Thai massage, Thai massage with pure coconut oil, Thai massage with oil mixed with Snake fruit extract, Control, Facial mask with Snake fruit extract, Control jelly, Jelly with Snake fruit juice
- Study 2: Facial mask with Snake fruit extract (Experimental): Participants were randomized to receive an arm. In this arm, participants received home-based program facial mask with Snake fruit extract for 30 min/day, 2 days/week for 12 weeks.
  Interventions: Other: Thai massage, Thai massage with pure coconut oil, Thai massage with oil mixed with Snake fruit extract, Control, Facial mask with Snake fruit extract, Control jelly, Jelly with Snake fruit juice
- Study 3: Control jelly (Active Comparator): Participants were randomized to receive an arm. In this arm, participants consumed with control jelly at 3.5 g/kg body weight. Consumption was taken at Burapha University.
  Interventions: Other: Thai massage, Thai massage with pure coconut oil, Thai massage with oil mixed with Snake fruit extract, Control, Facial mask with Snake fruit extract, Control jelly, Jelly with Snake fruit juice
- Study 3: Jelly with Snake fruit juice (Experimental): Participants were randomized to receive an arm. In this arm, participants consumed with jelly with Snake fruit juice at 3.5 g/kg body weight. Consumption was taken at Burapha University.
  Interventions: Other: Thai massage, Thai massage with pure coconut oil, Thai massage with oil mixed with Snake fruit extract, Control, Facial mask with Snake fruit extract, Control jelly, Jelly with Snake fruit juice

INTERVENTIONS:
Other: Thai massage, Thai massage with pure coconut oil, Thai massage with oil mixed with Snake fruit extract, Control, Facial mask with Snake fruit extract, Control jelly, Jelly with Snake fruit juice — Interventions among the 3 studies were categorized as other.

SUMMARY:
This study consisted of three sub-studies including 1) development and evaluation of body massage oil from Snake fruit on skin moisture, elasticity, oiliness, and melanin in healthy participants 2) development and evaluation of facial mask from Snake fruit on skin moisture, elasticity, oiliness, and melanin in healthy participants and 3) development and evaluation of ready-to-drink jelly from Snake fruit on controlling blood glucose and endurance time in healthy participants.

DETAILED DESCRIPTION:
Study 1: senventy-one male and female participants, aged 23.99 ± 5.68 years were randomly assigned into 3 groups including 1) control group (n = 23): participants received Thai massage without any oil for 1 hour/day, 1 day/week for 12 weeks 2) treatment-1 group (n = 23): participants received Thai massage with pure coconut oil which is a popular oil used in spa for 1 hour/day, 1 day/week for 12 weeks and 3) treatment-2 group (n = 25): participants received Thai massage with oil mixed with Snake fruit extract for 1 hour/day, 1 day/week for 12 weeks.

Study 2: fifty-nine male and female participants, aged 23.39 ± 4.84 years were randomly assigned into 2 groups including 1) control group (n = 29): participants did not receive any facial mask for 12 weeks and 2) treatment group (n = 30): participants received home-based program facial mask with Snake fruit extract for 30 min/day, 2 days/week for 12 weeks.

Study 3: this study was divided into 2 sub-stidies. Study 3.1: twenty-five male and female participants, aged 22.60 ± 3.33 years were randomly consumed with either control jelly or jelly with Snake fruit juice at 3.5 g/kg body weight. All participants were analyzed for blood glucose level before consumption and after consumption at 30, 60, 90, and 120 min. Study 3.2: twenty-three male and female participants, aged 21.57 ± 1.88 years were randomly consumed with either control jelly or jelly with Snake fruit juice at 3.5 g/kg body weight. After each consumption, all participants performed leg cycling at intensity 60% of maximal oxygen consumption as long as tolerance (time to exhaustion test).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Aged between 18 to 35 years
* Healthy
* Interested in body massage with oil or facial mask or jelly from Snake fruit

Exclusion Criteria:

* History of adverse effects from body massage
* Skin allergy
* Skin disorders
* Skin wounds
* History of allergy to coconut or plant oil
* History of allergy to facial mask, i.e., mask from fruit
* History of allergy to Snake fruit or gelatin
* Signs or symptoms of fever or infection
* Abnormal body mass index
* Regular smokers or alcohol drinkers (>2 times per week)
* Regular exerciser (>2 times per week or >150 min per week)
* Regular intake of dietary supplements, i.e., vitamins, antioxidants
* Hypertension, diabetes, cardiovascular disease, respiratory disease, endocrine disease, neuromuscular disease, musculoskeletal disease, liver disease, renal disease, immune disease, infectious disease, or cancer

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Level of skin moisture | Before intervention, immediately after intervention, ends of week 4, week 8, and week 12
  Study 1 and 2 determined level of skin moisture in arbitrary unit (no unit) using Multiprobe Adapter System with Corneometer® CM 825 probe
Level of skin elasticity | Before intervention, immediately after intervention, ends of week 4, week 8, and week 12
  Study 1 and 2 determined level of skin elasticity in arbitrary unit (no unit) using Multiprobe Adapter System with Cutometer® 580 probe
Level of skin oiliness | Before intervention, immediately after intervention, ends of week 4, week 8, and week 12
  Study 1 and 2 determined level of skin oiliness in arbitrary unit (no unit) using Multiprobe Adapter System with Sebumeter® SM 815 probe
Level of skin melanin | Before intervention, immediately after intervention, ends of week 4, week 8, and week 12
  Study 1 and 2 determined level of skin melanin in arbitrary unit (no unit) using Multiprobe Adapter System with Mexameter® MX18 probe
Level of blood glucose | Before jelly consumption and after jelly consumption at 30, 60, 90, and 120 minutes
  Study 3.1 determined level of blood glucose in mg/dL unit
Endurance time | After jelly consumption for 30 minutes
  Study 3.2 determined endurance time by cycling at 60% of maximum oxygen consumption as long as possible (time to exhaustion test)
Concentration of interferon-gamma | Before and immediately after endurance time test
  Study 3.2 determined concentration of interferon-gamma in serum in pg (picogram)/mL unit
Concentration of tumor necrosis factor-alpha | Before and immediately after endurance time test
  Study 3.2 determined concentration of tumor necrosis factor-alpha in serum in pg (picogram)/mL unit

CONTACTS AND LOCATIONS:
Overall Officials: Piyapong Prasertsri, Ph.D., Principal Investigator — Burapha University
Locations (1):
- Faculty of Allied Health Sciences, Burapha University, Mueang, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Boonla O, Chancharoen P, Padkao T, Teethaisong Y, Tangwattanachuleeporn M, Koowattanatianchai S, Prasertsri P. Acute ingestion of snake fruit jelly improves glycemic response, enhances endurance performance and antioxidant defense, and reduces inflammatory markers in healthy adults. J Int Soc Sports Nutr. 2025 Dec;22(1):2579029. doi: 10.1080/15502783.2025.2579029. Epub 2025 Oct 26. PMID 41139389